CLINICAL TRIAL: NCT00841828
Title: A Multicentre, Randomised Phase II to Compare Epirubicin (E) & Cyclophosphamide (C) Treatment Plus Docetaxel (D) & Trastuzumab vs. E & C Treatment Plus D & Lapatinib in Women With Primary Resectable or Locally Advanced HER2+ Breast Cancer
Brief Title: Trastuzumab Versus Lapatinib as Neoadjuvant Treatment for Her2+ Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2006-14; 2007-007031-13 (EudraCT Number)
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; Lapatinib; Neoadjuvant; Trastuzumab; Biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Epirubicin + Cyclophosphamide -> Docetaxel + Lapatinib
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Lapatinib
- Control (Active Comparator): Epirubicin + Cyclophosphamide -> Docetaxel + Trastuzumab
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Epirubicin
  Other Names: Ellence; Pharmorubicin
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar; Endoxan
Drug: Docetaxel
  Other Names: Taxotere
Drug: Lapatinib
  Other Names: Tykerb
  Arms: Experimental
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Control

SUMMARY:
Phase II randomized multicenter trial to compare Epirubicin and Cyclophosphamide plus Docetaxel and Trastuzumab with Epirubicin and Cyclophosphamide plus Docetaxel and Lapatinib for patients with positive HER2 and resectable or locally advanced breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, open label, randomized phase II trial. Women with primary cancer and overexpression of Human Epidermal Growth Factor Receptor 2 (HER2) who have not received prior treatment for invasive breast cancer will be included. The study will analyze the efficacy and tolerance of Lapatinib and Docetaxel and the Trastuzumab and Docetaxel after 4 cycles of Epirubicin and Cyclophosphamide in patients with breast cancer HER2 positive.

102 patients will be stratified according to tumor size and estrogen receptor status (positive or negative) to be randomized to receive one of the following treatment arms:

* Experimental arm: Epirubicin 90mg/m2 in combination with cyclophosphamide 600mg/m2 intravenous (IV) every 21 days for 4 cycles, followed by oral Lapatinib 1250mg once a day plus docetaxel 100mg/m2 IV every 21 days for 4 cycles with the administration of granulocyte-colony stimulating factor (G-CSF) between days 2 and 7 or on day +1 according to the G-CSF used by the site.
* Control arm: Epirubicin 90mg/m2 in combination with cyclophosphamide 600mg/m2 IV every 21 days for 4 cycles, followed by a loading dose of Trastuzumab 8mg/kg IV followed by Trastuzumab 6mg/kg IV every 3 weeks plus docetaxel 100mg/m2 IV every 21 days for 4 cycles with the administration of G-CSF between days 2 and 7 or on day +1 according to the G-CSF used by the site.

Treatment duration: The patients will be in treatment for an average of 6 months for both arms.

Study population: Patients with operable or locally advanced breast cancer, HER2 positive who are candidates to receive neoadjuvant treatment and who have not received pre-treatment for invasive breast cancer.

Population in study and number total of patients:

The aim is to determine if neoadjuvant treatment with selective therapy can increase the complete pathological response (pCR) in breast cancer by the determination of molecular markers in the tumoral sample before treatment. Then, and between 3 and 4 weeks after the last administration of Docetaxel, and 24 hours after the administration of Lapatinib, surgery will be performed and in the surgical sample will be determined the molecular markers analyzed before of the treatment in the tumor sample.

Patients with HER2 positive, defined as immunohistochemistry 3+ or positive fluorescence in situ hybridization (FISH), will be included. If immunohistochemistry 2+ it will be necessary to confirm the HER2 positive status by FISH. All results will be reevaluated later in the central laboratory.

Statistical consideration: The sample size has been calculated using the 2-stage Simon method and with pathological complete response (pCR) as the primary study end point. Sample size has been based on the null hypothesis of a pCR of 40% and an alternative hypothesis of a pCR of 60%. Assuming an alpha error of 0.05 and a test power of 80%, 92 evaluable patients will be required to be recruited and retained in the study. Sixteen patients per arm will be included in the first stage, for at least eight pCR per arm to be seen, and 30 additional patients per arm will be included in the second stage for a total of 46 evaluable patients in each arm. Assuming a 10% drop-out rate, 102 patients will be recruited.

The objective of the random distribution to treatment arms is to select the most active arm for a subsequent development. It is based on a standard of pCR of 40%, in order to detect an increase in the pCR rate of 60% in both arms, it would be necessary to include 46 patients in each arm (Simon's method in 2 stages (Optimal design)). It has been considered an error a = 0.05 and a power 80% statistics. Therefore, in the first stage it would be necessary to include 16 patients in each arm if we found more than 7 patients with pCR in each arm we will continue including until reaching the 46 in each arm. The results will be significant if we find at least 23 patients with pCR in each arm. Assuming that 10% of patients are not evaluable, the number The total number of patients to be included is 102 patients (51 patients per arm of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the written informed consent.
2. Histological documentation of breast cancer.
3. Stage I (T1, N0M0), IIA (T2N0M0); IIB (T2N1M0, T3N0M0), IIIA (TXN2M0) and IIIB (T3N1M0, T4NXM0) primary resectable breast cancer or locally advanced breast cancer.
4. HER2-positive breast cancer, defined as immunohistochemistry (IHQ) 3+ or positive FISH. When IHQ 2+ HER2 status must be assessed by FISH.
5. The patient granted her consent for taking a biopsy before treatment
6. The patient granted her consent for sending two tumor samples to central laboratory for molecular sub study.
7. Two weeks prior randomization pregnancy test negative for women of childbearing potential.
8. Women of childbearing potential must use adequate contraceptive measures during participation into study. Oral, injectable or implant hormonal contraceptives measure are not permitted.
9. A World Health Organization (WHO) performance status of 0 or 1 (Karnofsky ≥ 80)
10. Age > 18 years.
11. Absence of metastases disease
12. Baseline Electrocardiography (EKG) 12 weeks prior to randomization. Baseline left ventricular ejection fraction (LVEF) value within limit of normal value for the institution or > 50% of basal value
13. Normal laboratory test 2 weeks prior to randomization:

    Haematology values: Neutrophil count ≥ 1,5 x109/l; Platelets ≥ 100 x 109/l; Haemoglobin ≥ 10mg/dl Biochemistry values: serum total bilirubin ≤ 1 x Upper Limit of Normal (ULN); Aspartate aminotransferase (AST) (SGOT) and Alanine aminotransferase (ALT) (SGPT) ≤ 2,5 x ULN; alkaline phosphatase ≤ 5 x ULN. Patients which AST and/or ALT value are > 1,5 x ULN along with alkaline phosphatase value > 2,5 x ULN will be not included into the study.

    Renal function: serum creatinine ≤ 175 µmol/l (2 mg/dl). If the value is borderline, clearance creatinine must be ≥ 60 ml/min
14. 12 weeks prior to randomization the following assessments and procedures must be fulfilled: Bilateral mammography; Magnetic resonance imaging (MRI) Breast and axillary; Chest X-Ray (posterioanterior and lateral); Abdominal ultrasound; Chest CT-Scan; Abdominal CT-Scan. Bone Scan (if applicable)
15. Patients must be accessible for treatment and follow up

Exclusion Criteria:

1. Patients with lumpectomy, partial mastectomy, modified radical mastectomy are not allowed to include into study.
2. Prior Immunotherapy, hormonal therapy and chemotherapy for breast cancer is not allowed.
3. Prior therapy with anthracycline and taxanes (paclitaxel and docetaxel) is not permitted for any neoplasia.
4. Prior radiotherapy for breast cancer.
5. Bilateral invasive breast carcinoma
6. Pregnant or nursing patients. Negative pregnant test (serum or urine) 14 days prior to randomization.
7. HER 2 negative breast cancer
8. Patients of childbearing potential must be use adequate contraceptive measures during study treatment. No hormonal contraceptive measure is permitted.
9. Any M1 breast cancer
10. Any motor or sensorial neurotoxicity grade ≥ 2 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
11. Serious cardiac illness or medical conditions: Congestive heart failure, angina pectoris requiring specific treatment, myocardial infarction 1 year prior to enroll in the study; poorly controlled hypertension or high-risk uncontrolled arrhythmias.

    History of significative neurological or psychiatric disease (psychotic, dementia or attack) what is unable to patient to grant her informed consent.

    Uncontrolled severe Infection Uncontrolled diabetes mellitus, active peptic ulcer
12. Current malignancy or previous malignancy other that breast cancer. Exception cell carcinoma of the skin no melanoma, carcinoma in situ of the cervix or any other cancer in the past 10 years.
13. Long term treatment with corticoids except 6 months prior to inclusion in the study and low doses (≤ 20 mg methylprednisolone or equivalent)
14. Corticoid use contraindication
15. Concomitant hormonal replacement therapy. Previous treatment should be interrupted before inclusion into study.
16. Cardiopathy what stops patient taking Docetaxel and Trastuzumab: myocardial infarction recorded; angina pectoris requiring specific treatment; any congestive heart failure recorded; arrhythmia grade 3 or 4 according to NCI CTCAE version 3; any relevant valvular disease; chest X ray which shows cardiomegaly or EKG which shows ventricular hypertrophy unless LVEF value has been ≥ lower normal limit in the last 3 months.
17. Poorly controlled hypertension (systolic > 180 mm Hg or diastolic > 100 mm Hg). The patients with controlled hypertension under treatment can be included into study
18. Patients under treatment of arrhythmia, angina or congestive heart failure with drug which modifies cardiac conduction (after digital, beta blocker or inhibitors calcium channel) are excluded. However if these drugs are took for arterial tension the patient can be included into study.
19. The patient must interrupt concomitant treatment with hormonal therapy ej. raloxifene, tamoxifen and selective estrogen receptor modulators (SERM) prior to randomization.
20. Concomitant use of inhibitors and inductors of enzyme CYP3A4 complex (ketoconazole, itraconazole or grape juice; rifampicin, carbamazepin or fenitoin) are not permitted. Also, drug are substrate of enzyme CYP2C8 complex is not permitted along with lapatinib treatment.
21. Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial within 30 days prior to randomization into study.
22. Concomitant treatment with other anticancer therapy
23. Hypersensitivity reaction to drugs trastuzumab, lapatinib or their excipients.
24. Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Clínico Universitario de Valencia; Study Director, Study Director — Hospital Clínico Universitario Virgen de la Victoria; Study Director, Study Director — Hospital del Mar
Locations (26):
- Spain (26):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Xarxa Asistencial de Manresa, Manresa, Barcelona
  - Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital del Espíritu Santo, Santa Coloma de Gramenet, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Xeral Cíes, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Yagüe, Burgos
  - Complejo Hospitalario San Pedro de Alcántara, Cáceres
  - Complejo Hospitalario Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Alba E, Albanell J, de la Haba J, Barnadas A, Calvo L, Sanchez-Rovira P, Ramos M, Rojo F, Burgues O, Carrasco E, Caballero R, Porras I, Tibau A, Camara MC, Lluch A. Trastuzumab or lapatinib with standard chemotherapy for HER2-positive breast cancer: results from the GEICAM/2006-14 trial. Br J Cancer. 2014 Mar 4;110(5):1139-47. doi: 10.1038/bjc.2013.831. Epub 2014 Jan 23. PMID 24457911
- See also: Sponsor's website — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: EC -> D + Lapatinib: EC -> D + Lapatinib
  Drugs plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles -> Docetaxel + Lapatinib each 21 days for 4 cycles
- Arm 2: EC -> D + Trastuzumab: EC -> D + Trastuzumab
  Drug plus Biological
  EC each 21 days for 4 cycles -> Docetaxel + Trastuzumab each 21 days for 4 cycles
Period: Overall Study
Arm/Group | Arm 1: EC -> D + Lapatinib | Arm 2: EC -> D + Trastuzumab
Started | 52 | 50
Completed | 42 | 48
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: EC -> D + Lapatinib: Epirubicin and Cyclophosphamide (EC) followed by Docetaxel (D) and Lapatinib
  Drugs plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles followed by Docetaxel and Lapatinib each 21 days for 4 cycles
- Arm 2: EC -> D + Trastuzumab: Epirubicin and Cyclophosphamide (EC) followed by Docetaxel (D) and Trastuzumab
  Drug plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles followed by Docetaxel and Trastuzumab each 21 days for 4 cycles
- Total: Total of all reporting groups
Arm/Group | Arm 1: EC -> D + Lapatinib | Arm 2: EC -> D + Trastuzumab | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Median (Full Range); unit: years] | 48 [30 to 79] | 48.5 [32 to 74] | 48 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 52 | 50 | 102
Menopausal Status [Number; unit: participants]
  Premenopausal | 28 | 29 | 57
  Postmenopausal | 24 | 21 | 45
Estrogen Receptor [Number; unit: participants]
  Positive | 29 | 30 | 59
  Negative | 23 | 20 | 43
Tumor Size [Median (Full Range); unit: centimeters] | 3.5 [1 to 15.8] | 3.3 [1 to 10] | 3.3 [1 to 15.8]
Nodal Status [Number; unit: participants]
  N0=no regional lymph node metastases | 19 | 13 | 32
  N1=metastases 1-3 axillary lymph node/s | 32 | 35 | 67
  N2=metastases in 4-9 axillary lymph nodes | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathological Response (pCR) Rate in Breast and Axilla According to the Miller&Payne Criteria (G5-A and G5-D).
Description: Within 3-4 weeks after last docetaxel dose the surgery was performed to evaluate pathological response. According to the Miller&Payne Criteria, pCR in node-negative patients is a grade 5-A and in node-positive patients is a grade 5-D.
Time Frame: Up to 16 weeks
Population: Arm 1: 1 patient not included in this analysis due to negative Fluorescence in situ hybridization (FISH) result.
  Arm 2: 2 patients not included in this analysis due to negative Fluorescence in situ hybridization (FISH) result.
Measure: Number (95% Confidence Interval); unit: percentage of participants with pCR
Groups:
- Arm 1: EC -> D + Lapatinib: EC -> D + Lapatinib
  Drugs plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles -> Docetaxel (D) + lapatinib each 21 days for 4 cycles)
- Arm 2: EC -> D + Trastuzumab: EC -> D + Trastuzumab
  Drug plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles -> Docetaxel (D) + Trastuzumab each 21 days for 4 cycles
Arm/Group | Arm 1: EC -> D + Lapatinib | Arm 2: EC -> D + Trastuzumab
Number analyzed (Participants) | 51 | 48
percentage of participants with pCR | 23.5 [11.9 to 35.1] | 47.9 [33.8 to 62.0]

2. Secondary Outcome: Overall Clinical Response Rate (ORR)
Description: Overall clinical response was evaluated according to the Response Evaluation Criteria in Solid Tumours (RECIST) criteria (Therasse et al, 2000). Is defined as the sum of Complete responses plus Partial responses.
  It was evaluated after the fourth EC cycle and before surgery using ultrasound, mammography, or MRI.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm 1: EC -> D + Lapatinib: EC -> D + Lapatinib
  Drugs plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles -> Docetaxel (D) + lapatinib each 21 days for 4 cycles
- Arm 2: EC -> D + Trastuzumab: EC -> D + Trastuzumab
  Drug plus Biological
  Epirubicin + Cyclophosphamide (EC) each 21 days for 4 cycles -> Docetaxel + Trastuzumab each 21 days for 4 cycles
Arm/Group | Arm 1: EC -> D + Lapatinib | Arm 2: EC -> D + Trastuzumab
Number analyzed (Participants) | 51 | 48
percentage of participants | 62.7 [49.4 to 76] | 77.1 [65.2 to 89]

ADVERSE EVENTS:
Time Frame: Through study treatment up to 24 week
Description: These Adverse Events are by patient (not per cycle). Only grades 3 and 4 are specified.
Arm/Group | Arm 1: EC -> D + Lapatinib | Arm 2: EC -> D + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 11/52 | 4/50
Other Adverse Events (participants affected / at risk) | 28/52 | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: EC -> D + Lapatinib (N=52) | Arm 2: EC -> D + Trastuzumab (N=50)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: EC -> D + Lapatinib (N=52) | Arm 2: EC -> D + Trastuzumab (N=50)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10 (10) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 13 (13) | 10 (10)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
ALT, SGPT (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No